CLINICAL TRIAL: NCT02235948
Title: Efficacy and Safety of Folic Acid Supplementation Lowering Arsenic in a Chronic, Low-level Exposed Arsenic Population: a Randomized, Double-blind, Placebo Controlled Clinical Trial.
Brief Title: Effects of Folic Acid Supplementation on Arsenic Lowering
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiao Xiao, MD, PhD, professor, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Y211045
Record Dates: First submitted 2014-08-28; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Arsenic Poisoning; Toxic Effect of Arsenic and Its Compounds
Keywords: arsenic induced health problem; modifying effects; folic acid; oxidative damage; clinical trial
MeSH Terms: conditions — Arsenic Poisoning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- folic acid (Experimental): folic acid supplementation placebo controlled
  Interventions: Drug: folic acid supplementation

INTERVENTIONS:
Drug: folic acid supplementation — 0.8mg folic acid/day
  Other Names: placebo controlled

SUMMARY:
The purpose of this study is to determine whether folic acid supplementation are effective on arsenic lowering in a chronic, low-level arsenic exposed population.

DETAILED DESCRIPTION:
Outcome measure:

Changes of arsenic metabolites at baseline and week 8

Methods High-performance liquid chromatography (HPLC)

ELIGIBILITY:
Inclusion Criteria:

* Men or women more than 18 years of age and chronically exposed to arsenic (arsenic concentration of the drinking water >10ug/L);
* Population who had no folic acid supplementation in the 2 weeks before the study;
* Women of childbearing age agreed to use a reliable contraception method during the study;
* Everyone volunteered to participate and signed informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding women;
* Allergic to folic acid;
* Having clearly defined allergic history;
* Reported long-term use of folic acid and other vitamins B;
* Having obvious signs or laboratory abnormalities which could affect the efficacy of folic acid;
* Unsuitable to participate in the study based on the judgment of the investigators;
* Not agree to cancel the medications which may affect serum folate concentration during the study period;
* Subjects who plan to become pregnant during the study or move out of the area within the study period;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of urine arsenic metabolites between baseline and week 8 | baseline, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Xiao, MD, PhD, Study Director — Wenzhou Medical University

REFERENCES:
- [Derived] Bae S, Kamynina E, Guetterman HM, Farinola AF, Caudill MA, Berry RJ, Cassano PA, Stover PJ. Provision of folic acid for reducing arsenic toxicity in arsenic-exposed children and adults. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD012649. doi: 10.1002/14651858.CD012649.pub2. PMID 34661903
- [Derived] Wei Y, Jia C, Lan Y, Hou X, Zuo J, Li J, Wang T, Mao G. The association of tryptophan and phenylalanine are associated with arsenic-induced skin lesions in a Chinese population chronically exposed to arsenic via drinking water: a case-control study. BMJ Open. 2019 Oct 30;9(10):e025336. doi: 10.1136/bmjopen-2018-025336. PMID 31666259
- [Derived] Guo X, Cui H, Zhang H, Guan X, Zhang Z, Jia C, Wu J, Yang H, Qiu W, Zhang C, Yang Z, Chen Z, Mao G. Protective Effect of Folic Acid on Oxidative DNA Damage: A Randomized, Double-Blind, and Placebo Controlled Clinical Trial. Medicine (Baltimore). 2015 Nov;94(45):e1872. doi: 10.1097/MD.0000000000001872. PMID 26559255